CLINICAL TRIAL: NCT06762678
Title: Transcriptomic Approach for the Identification and Prioritization of Genome Variants in Neurodevelopmental Disorders With Malformation
Acronym: ATOMICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC23_0426; 2024-A01997-40 (Other: ANSM)
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Neurodevelopmental Disorders and Developmental Abnormalities
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNA sequencing and trio whole genome sequencing (Other): Each index case will be analysed through RNA sequencing and trio whole genome sequencing. The biologists in charge of data interpretation in this arm will have access to every data.
  Interventions: Diagnostic Test: RNA sequencing and whole genome sequencing in a trio way
- Genome sequencing trio only (Other): Each index case will be analysed through RNA sequencing and trio whole genome sequencing. In this arm however, the biologists in charge of data interpretation will be blinded from RNA sequencing results
  Interventions: Diagnostic Test: RNA sequencing and whole genome sequencing in a trio way

INTERVENTIONS:
Diagnostic Test: RNA sequencing and whole genome sequencing in a trio way — Patient is not required to be blinded

SUMMARY:
Three million persons in France are impacted by rare diseases. Amid the 7000 different diseases which are identified today, neurodevelopmental disorders are the main symptoms found interesting 35 000 birth every years, according to the French Health Authority. In half of these cases, patients are under 5 years old and a molecular diagnosis is only available in 50% of them, associated with a diagnostic wandering exceeding 5 years for 25% of every patients.

High throughput DNA sequencing technologies are powerful tools to elucidate new causative variants. Although the diagnostic yield was refined by DNA-seq, data interpretation and technology limits remain the two major obstacles which still need be overcame. Missing a molecular diagnosis through a genomic approach alone highlight the need to integrate multi-omic approaches such as Ribonucleic Acid sequencing. This sequencing level allows new insight such like the evidence of aberrant gene expression, mono allelic allele expression, or abnormal alternative splicing. It makes possible too, to detect variants which are unable to be found via genome sequencing only.

Recently, a diagnostic performance improvement has been described trough the association of the two technics, i.e. Ribonucleic Acid-seq and genome sequencing, in a context of neuromuscular diseases. However, only few studies were carry out on neurodevelopmental disorders in addition with malformative features. We demonstrated by the end of 2022, a diagnostic results enhancement by carrying genome sequencing plus Ribonucleic Acid-seq at the same time on patient with previously exome negative analysis. Moreover in 2023, Dekker et al. work shed light on a diagnostic yield improvement via the same analytic schema.

In face of those first observations, our study aims to evaluate the diagnostic contribution of Ribonucleic Acid-seq paired with genome sequencing in a trio way versus the genome sequencing in a solo way, to identify the find a final diagnosis for patient presenting neurodevelopmental disorders with developmental abnormalities and without an evident diagnosis after chromosome microarray and/or exome sequencing analysis.

To successfully carry out our study, we plan to recruit patient in a protocol considered with minimal risk and minimal constraints, to compare Ribonucleic Acid-seq performed on fibroblasts, in addition to genome sequencing in a solo or a trio manner, to trio genome sequencing alone, with the final objective in mind to obtain an etiology diagnostic for a patient presenting with neurodevelopmental disorders and development abnormalities.

ELIGIBILITY:
Inclusion Criteria :

* children or adult without any age limit, with neurodevelopmental disorders defined by :
* between 0 and 5 years old with severe developmental delays regarding motor and/or language acquisitions, and/or social communication disorders,
* > 6 years old with intellectual deficiency whatever the severity (with if available, neuropsychological evaluation), with potential associated manifestations such as epilepsy and/or autism, and/or behaviour troubles and/or attention deficit hyperactivity disorder ;
* with developmental anomalies and/or dimorphism ;
* without any evidence of clinical diagnosis
* negative chromosomal microarray and/or exome sequencing
* negative fragile X syndrome
* skin biopsy feasible or RNA sample extracted from fibroblast culture, available to be used in a research context inside the lab center
* consent obtained from the participant or, consent from legal representatives for a minor patient or a patient unable to consent
* participant affiliated to the french security regimen or equivalent

Exclusion Criteria:

* Neurodevelopmental disorders with developmental anomaly from non genetic causes or highly evident diagnosis for which a molecular test is available in routine practices and whose the cost is inferior than the cost of the genome and the RNA sequencing
* unwillingness to participate, from the patient or from the legal representatives
* Pregnant or lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Compare the interest of RNA sequencing in addition to a genome sequencing in trio, versus a genome sequencing trio analyse carried out alone, to identify the etiologic diagnosis of patient with neurodevelopmental disorders and developmental abnormalities | 12 months
  To compare the interest of RNA sequencing, carried out into fibroblasts in addition to a genome sequencing in trio, versus a genome sequencing-trio analyse carried out alone, to identify the etiologic diagnosis of patient with neurodevelopmental disorders and developmental abnormalities, without any obvious clinical diagnosis a priori, and without no identified result after Chromosomal Microarray and/or solo or trio exome sequencing Number of class 4 or class 5 (according the American College of Medical Genetics classification) variants newly identified and allowing a diagnosis to explain patient' symptoms, following RNA sequencing + genome sequencing-trio, vs genome sequencing trio alone.

IPD SHARING:
Plan to Share IPD: Undecided